CLINICAL TRIAL: NCT07300852
Title: The Effectiveness of DSLT in Asian Normal Tension Glaucoma Patients
Brief Title: DSLT in Normal Tension Glaucoma (NTG) Asian Eyes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ngoc Nguyen Inc. (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Ngoc Nguyen M.D., Principal Investigator, Ngoc Nguyen Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTG_DSLT-001
Record Dates: First submitted 2025-12-09; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Normal Tension Glaucoma (NTG); Glaucoma; Open Angle Glaucoma (OAG); Glaucoma, Open Angle
Keywords: DSLT; Direct Selective Laser Trabeculoplasty; NTG; Glaucoma; Normal Tension Glaucoma; BELKIN Vision Eagle; Glaucoma laser treatment; Asian glaucoma; Intraocular pressure; SLT alternative; Glaucoma medications reduction
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DSLT Treatment Arm (Experimental): Participants will receive Direct Selective Laser Trabeculoplasty (DSLT) using the BELKIN Vision Eagle device. The procedure is performed without a contact lens and delivers non-contact laser energy to the trabecular meshwork to lower intraocular pressure. All participants undergo standard pre- and post-procedure evaluations, including IOP measurements, visual field testing, and OCT imaging.
  Interventions: Device: Direct Selective Laser Trabeculoplasty (DSLT)

INTERVENTIONS:
Device: Direct Selective Laser Trabeculoplasty (DSLT) — Direct Selective Laser Trabeculoplasty (DSLT) is a non-contact laser procedure that delivers energy to the trabecular meshwork without the need for a gonioscopy lens. The BELKIN Vision Eagle device automatically aligns and applies laser pulses to lower intraocular pressure in subjects with normal tension glaucoma. All participants receive a single DSLT treatment followed by routine post-procedure evaluations including IOP checks, visual field testing, and OCT imaging.
  Other Names: BELKIN Vision Eagle; Non-contact SLT; DSLT Laser Treatment; Direct Selective Laser Trabeculoplasty

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of direct selective laser trabeculoplasty (DSLT) or laser treatment in Asian patients with normal tension glaucoma. The main question it aims to answer is:

Does the DSLT reduce intraocular pressure (IOP) and medication use in Asian NTG subjects? Participants will attend routine follow-up visits with their eye surgeon and glaucoma testing such as optical coherence tomography (OCT) imaging and visual field test(s) after the laser study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Asian descent
* NTG diagnosis: glaucomatous optic neuropathy in patients with IOP measurements consistently lower than 21 mmHg
* Mean deviation (MD) of the visual field between 0 to -12dB
* No significant central vision loss within 5 degrees within 5th percentile
* Age ≥20 years
* NTG patients who are medically controlled on 1-3 medications and safe to wash out or IOP is still insufficient from medications and safe to washout
* Shaffer grade II or more on 3 of the 4 quadrants
* Central corneal thickness (CCT) 450-600µm
* All participants are able to provide written informed consent before participation

Exclusion Criteria:

* Angle closure glaucoma or narrow angle status post laser peripheral iridotomy (LPI), or any other open angle glaucoma excluding NTG
* History of SLT within last 2 years
* History intraocular surgery including refractive surgery, except for history of cataract surgery that has been greater than 1 year
* Patients anticipating cataract surgery during the study follow-up period
* Unable to have DSLT procedure due to pre-limbal findings
* Any presence of relevant ocular diseases including retinal disease with no confirmed cure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) | 12 months post procedure
  Absolute change in washed-out intraocular pressure (IOP) at 12 months compared to washed-out baseline IOP. Following a 6-week washout at baseline and again at month 11, IOP will be measured using standard tonometry to assess the effect of Direct Selective Laser Trabeculoplasty (DSLT) on pressure reduction.

SECONDARY OUTCOMES:
Number of Glaucoma Medications Reduced | 12 months post-procedure
  Change in the number of topical glaucoma medications required to control intraocular pressure at 11 months compared to baseline, to evaluate whether DSLT decreases medication burden.
Proportion of Patients Who Are Medication-Free | 12 months post-procedure
  Proportion of participants who require zero topical glaucoma medications at 11 months after DSLT treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ngoc Nguyen M.D., San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) for this study. The sample size is small and sharing de-identified datasets may not adequately protect participant privacy.

DOCUMENTS (2):
  • Study Protocol (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT07300852/Prot_000.pdf
  • Informed Consent Form (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT07300852/ICF_001.pdf